CLINICAL TRIAL: NCT00193258
Title: A Phase I/II Trial of Bevacizumab (Avastin), Erlotinib (Tarceva), and Imatinib (Gleevec) in the Treatment of Patients With Advanced Renal Cell Carcinoma
Brief Title: Bevacizumab, Erlotinib, and Imatinib in the Treatment of Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 22
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Recurrent clear cell renal cell carcinoma; Bevacizumab; Erlotinib; Imatinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Erlotinib Hydrochloride; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): In the phase I portion:
  Bevacizumab 10 mg/kg slow IV infusion on days 1 and 15 of each 28-day course
  Erlotinib 150 mg orally daily
  Imatinib 300 mg orally daily or 400 mg orally daily
  In the phase II portion:
  Bevacizumab 10 mg/kg 30-60 minute IV infusion on days 1 and 15 of every 28 day cycle
  Erlotinib 150 mg orally daily
  Imatinib 400 mg orally daily
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Imatinib

INTERVENTIONS:
Drug: Bevacizumab — 10mg/kg IV infusion every 2 weeks
  Other Names: Avastin
Drug: Erlotinib — 150 mg po daily
  Other Names: Tarceva
Drug: Imatinib — 400-600mg daily
  Other Names: STI571, Gleevec, Glivec, imatinib mesilate (INN)

SUMMARY:
This phase I/II trial will evaluate the bevacizumab/erlotinib combination with the addition of imatinib (Gleevec). The combined inhibition greatly enhances the anti-tumor effects. Although the safety of the bevacizumab/erlotinib/imatinib combination has not yet been demonstrated, the mild to moderate side effects of all of these agents are not predicted to cause prohibitive toxicity. A brief phase I portion will be included in this trial, to optimize doses of the 3 agents prior to proceeding with the phase II trial.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

Bevacizumab + Erlotinib + Imatinib

A brief phase I dose escalation study will be performed to define the imatinib dose that will be used.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic or unresectable clear cell renal carcinoma confirmed by biopsy
* Previous nephrectomy is required
* Maximum of 1 previous systemic regimen for metastatic disease.
* Able to perform activities of daily living with minimal assistance
* Measurable disease
* Adequate bone marrow, liver and kidney
* Written informed consent.

Exclusion Criteria:

* Age < 18 years
* Treatment with more than 1 previous systemic regimen
* History of heart attack within 6 months
* Clinically significant cardiovascular disease
* Moderate to severe vascular disease.
* Active brain metastases.
* History or evidence by physical examination of brain tumor
* Seizures not controlled with standard medical therapy
* history of stroke or other serious disorders of the nervous system
* Clinical history of coughing or vomiting blood within the past 3 months.
* PEG tubes or G tubes
* Chronic therapy with NSAIDS or other platelet inhibitors
* Proteinuria
* Nonhealing wound, ulcer, or long bone fracture
* Clinical evidence or history of a bleeding disorder
* Requiring full dose anticoagulation with coumadin
* Receiving chronic steroid therapy
* Significant medical conditions.
* Tumors other than clear cell
* History of stroke within 6 months.
* History of abdominal fistula,perforation,or abscess within 6 months.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2004-06; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Sosman JA, Burris HA 3rd, Farley C, Cucullu H, Yost K, Hart LL, Sylvester L, Waterhouse DM, Greco FA. Treatment of advanced renal cell carcinoma with the combination bevacizumab/erlotinib/imatinib: a phase I/II trial. Clin Genitourin Cancer. 2007 Dec;5(7):427-32. doi: 10.3816/CGC.2007.n.030. PMID 18272024
- See also: Published article in Clinical Genitourinary Cancer — http://cigjournals.metapress.com/content/78747811327l1q78/?p=add93b1605a842cb946ca178813c9b17&pi=2

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab/Erlotinib/Imatinib: In the phase I portion: Bevacizumab 10 mg/kg slow IV infusion on days 1 and 15 of each 28-day course Erlotinib 150 mg orally daily Imatinib 300 mg orally daily or 400 mg orally daily In the phase II portion: Bevacizumab 10 mg/kg 30-60 minute IV infusion on days 1 and 15 of every 28 day cycle Erlotinib 150 mg orally daily Imatinib 400 mg orally daily
Period: Overall Study
Arm/Group | Bevacizumab/Erlotinib/Imatinib
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab/Erlotinib/Imatinib
Number analyzed (Participants) | 94
Age Continuous [Median (Full Range); unit: years] | 60 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 74
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: Eighty-seven of 94 patients (93%) received ≥ 2 months of treatment and were fully evaluable for response. Seven patients discontinued treatment during the first 8 weeks. One of these 7 patients had evidence of rapid tumor progression, whereas the remaining 6 patients discontinued treatment because of toxicity or for personal reasons.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab/Erlotinib/Imatinib
Number analyzed (Participants) | 88
percentage of participants | 17 [9 to 26]

2. Primary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Time Frame: 18 months
Population: All patients enrolled in the trial
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Erlotinib/Imatinib
Number analyzed (Participants) | 94
months | 8.9 [6.6 to 10.9]

3. Primary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 24 months
Population: All patients enrolled in the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Erlotinib/Imatinib
Number analyzed (Participants) | 94
months | 17.2 [12.9 to 21]

ADVERSE EVENTS:
Arm/Group | Bevacizumab/Erlotinib/Imatinib
Serious Adverse Events (participants affected / at risk) | 45/94
Other Adverse Events (participants affected / at risk) | 83/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Erlotinib/Imatinib (N=94)
Hypertensive Emergency (Cardiac disorders) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1)
Acute Sepsis Syndrome (Infections and infestations) | 1 (1)
Large Pericetal Abscess (Gastrointestinal disorders) | 1 (1)
Severe Enteritis with likely bowel perforation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Spinal Cord compression (Nervous system disorders) | 1 (1)
Impending pathologic fracture of Right Proximal femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Superficial subcutaneous postoperative wound (Infections and infestations) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (3)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (2)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Wedge resection/biopsy of known nodule at left (Surgical and medical procedures) | 1 (1)
Choleocystitis (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Rt. pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subacute Infarct left posterior cerebral artery (Vascular disorders) | 1 (1)
GU obstruction (Gastrointestinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Renal Insufficiency (Renal and urinary disorders) | 1 (1)
CHF (Cardiac disorders) | 1 (1)
Wound Complication (Infections and infestations) | 1 (1)
Cardiac Ischemia (Cardiac disorders) | 1 (1)
Fecal Impaction (Gastrointestinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Intercranial Hemorrhage (Nervous system disorders) | 1 (1)
Hemoptysis (Gastrointestinal disorders) | 2 (3)
Gross Hematuria (Renal and urinary disorders) | 1 (2)
Duodenal Ulcer with Bleeding (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Erlotinib/Imatinib (N=94)
Allergic rhinitis (Immune system disorders) | 5 (26)
Hair Loss/Alopecia (Skin and subcutaneous tissue disorders) | 22 (72)
Anorexia (Gastrointestinal disorders) | 54 (187)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (33) — Arthralgia
Rigor/chills (General disorders) | 9 (16)
Constipation (Gastrointestinal disorders) | 22 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (60)
Cramps (abdominal) (Gastrointestinal disorders) | 8 (14)
Creatinine (Metabolism and nutrition disorders) | 5 (12)
Dehydration (Gastrointestinal disorders) | 12 (16)
Mood Alteration - Depression (Nervous system disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 83 (489)
Dizziness (Nervous system disorders) | 6 (10)
Heartburn/dyspepsia (Gastrointestinal disorders) | 14 (32)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (60)
Edema (Blood and lymphatic system disorders) | 29 (49)
Bleeding (Vascular disorders) | 30 (77)
Fatigue (General disorders) | 82 (424)
Fever (General disorders) | 15 (21)
Flatulence (Gastrointestinal disorders) | 10 (47)
Headache (Nervous system disorders) | 19 (33)
Hematuria (Renal and urinary disorders) | 15 (48)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (18)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 6 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (45)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypersensitivity (Immune system disorders) | 5 (9)
Hypertension (Cardiac disorders) | 21 (136)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (18)
Hyponatremia (Metabolism and nutrition disorders) | 7 (12)
Infection (Infections and infestations) | 43 (127)
Insomnia (General disorders) | 14 (45)
Mucositis (Gastrointestinal disorders) | 11 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (15)
Nausea (Gastrointestinal disorders) | 74 (198)
Neuropathy (Nervous system disorders) | 19 (59)
Pain (General disorders) | 18 (35)
Pain (abdominal) (Gastrointestinal disorders) | 6 (9)
Pain (back) (Musculoskeletal and connective tissue disorders) | 8 (21)
Proteinuria (Metabolism and nutrition disorders) | 69 (288)
Rash (Skin and subcutaneous tissue disorders) | 80 (517)
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Skin (dry) (Skin and subcutaneous tissue disorders) | 20 (75)
Skin (pruritis) (Skin and subcutaneous tissue disorders) | 14 (31)
Stomatitis (Gastrointestinal disorders) | 13 (25)
Taste change (Gastrointestinal disorders) | 5 (34)
Taste disturbance (Gastrointestinal disorders) | 36 (129)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (15)
Weight Loss (General disorders) | 27 (92)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 7 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.